CLINICAL TRIAL: NCT03245086
Title: Multi-center, Non-randomized Prospective Observation Study Comparing Ferguson Hemorrhoidectomy and Transanal Hemorrhoidal Dearterialization (THD) for Prolapsed, Nonincarcerated, Reducible Hemorrhoids in Terms of 1-year Recurrence
Brief Title: Multicenter Prospective Trial on Hemorrhoids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: THD America (Unknown)
Responsible Party: Principal Investigator, George Angelos, George Angelos, MD, MS, Stony Brook University
Other Study IDs: 934287
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Transanal hemorrhoid dearterialization (THD): Patients with prolapsed, non-incarcerated, reducible hemorrhoids in at least 3 columns undergoing transanal hemorrhoid dearterialization (THD).
  Interventions: Device: Transanal hemorrhoid dearterialization
- Ferguson hemorrhoidectomy: Patients with prolapsed, non-incarcerated, reducible hemorrhoids in at least 3 columns undergoing Ferguson hemorrhoidectomy.
  Interventions: Procedure: Ferguson hemorrhoidectomy

INTERVENTIONS:
Device: Transanal hemorrhoid dearterialization — The hemorrhoids are operated in their natural position and not distorted by eversion The proctoscope is fully introduced transanally to reach the lower rectum. Under Doppler guidance, six arterial signals are found circumferentially above the dentate line. The approach to make the 'dearterialization' involves the transfixation of the rectal mucosa and submucosa to entrap the artery using a suture. Mucopexy is performed after the artery ligation with the same suture used for the dearterialization. Finally, the suture is tied to fix the mucopexy.
  Other Names: THD
  Groups: Transanal hemorrhoid dearterialization (THD)
Procedure: Ferguson hemorrhoidectomy — The hemorrhoids are operated in their natural position and not distorted by eversion. A Ferguson-Hill retractor is used to expose the hemorrhoids. Dissection with scissors is directed up to the dentate line where the fibers of the sphincter muscles are exposed and only a mucosal pedicle remains attached. A Buie-Smith crushing clamp is applied to this pedicle and the hemorrhoidal mass is excised at the superior level of the clamp. The pedicle is then ligated and the crushing clamp is removed. After dissection of the intermuscular septum is complete, the margins of the wound are drawn upward into the anal canal with stitches and are secured to the pedicle by the same suture. The remainder of the wound is closed with a stitch tied at the outer extremity of the wound using the same suture.
  Groups: Ferguson hemorrhoidectomy

SUMMARY:
This study will compare Ferguson hemorrhoidectomy and THD in terms of one-year recurrence in a large population (N=492). Recurrence is defined as prolapsing internal hemorrhoids at physical examination performed by a colorectal surgeon.

DETAILED DESCRIPTION:
This is a multicenter, parallel arm, non-randomized prospective data collection trial comparing Ferguson hemorrhoidectomy and THD in terms of recurrence rates at one-year. All subjects will already be scheduled for either Ferguson or THD hemorrhoidectomy, the surgery is NOT part of the research. Although a randomized study would control for variation among surgeons, this study design provides the best patient safety since the surgeons will perform the technique they do most frequently. Variability in the patient population will be managed with a conservative sample size, which allows for a multivariate analysis of the sample populations if any confounding variables are noted during initial data analyses. In addition, the variability will be minimized with stringent and detailed inclusion/exclusion criteria in terms of hemorrhoidal disease. Patients will be enrolled and followed for one year. Participating surgeons will be credentialed and each participating surgeon will enroll up to ten consecutive patients.

The primary endpoint of this study is to compare Ferguson hemorrhoidectomy and THD in terms of recurrence rates at one-year. Recurrence is defined as prolapsing internal hemorrhoids at physical examination performed by a colorectal surgeon.

ELIGIBILITY:
Inclusion Criteria:

Patient must be:

* At least 18 years-old
* Able to sign informed consent
* Presenting with prolapsed, non-incarcerated, reducible hemorrhoids in at least 3 columns at physical examination and scheduled for either Ferguson or THD hemorrhoidectomy.

Exclusion Criteria:

* Any prior anorectal surgery except for conventional office-based interventions (rubber band ligation, sclerotherapy, and infrared coagulation)
* Prior pelvic radiotherapy
* Inflammatory bowel diseases
* Pre-existing fecal incontinence (Wexner score5 ≥8)
* Pre-existing chronic anal diseases
* Grades III and IV gynecological and obstetrical trauma per medical history and/or physical examination
* Connective tissue disorders
* Subject is pregnant
* Subject is under incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with prolapsed, non-incarcerated, reducible hemorrhoids in at least 3 columns at physical examination and scheduled for either Ferguson or THD hemorrhoidectomy.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Estimated)
Dates: Start 2016-08-17 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence rates | 1-year
  The primary endpoint of this study is to compare Ferguson hemorrhoidectomy and THD in terms of recurrence rates at one-year. Recurrence is defined as prolapsing internal hemorrhoids at physical examination performed by a colorectal surgeon.

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  The secondary outcomes include postoperative complications (i.e. urinary retention, constipation, dysuria, pruritis ani, anal pain, anal stenosis, unhealed wound, fissure, fecal urgency, incontinence- flatus, incontinence- stool)

CONTACTS AND LOCATIONS:
Overall Officials: George Angelos, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.

REFERENCES:
- [Background] FERGUSON JA, HEATON JR. Closed hemorrhoidectomy. Dis Colon Rectum. 1959 Mar-Apr;2(2):176-9. doi: 10.1007/BF02616713. No abstract available. PMID 13652788
- [Background] Ratto C, Parello A, Veronese E, Cudazzo E, D'Agostino E, Pagano C, Cavazzoni E, Brugnano L, Litta F. Doppler-guided transanal haemorrhoidal dearterialization for haemorrhoids: results from a multicentre trial. Colorectal Dis. 2015 Jan;17(1):O10-9. doi: 10.1111/codi.12779. PMID 25213152
- [Derived] Gachabayov M, Angelos G, George G, Kajmolli A, McGuirk M, Bergamaschi R. A Multicenter Prospective Non-Randomized Study Comparing Ferguson Hemorrhoidectomy and Transanal Hemorrhoidal Dearterialization for Prolapsed, Nonincarcerated, Reducible Hemorrhoids: A Study Protocol. Surg Technol Int. 2020 Nov 28;37:109-112. PMID 33238029